CLINICAL TRIAL: NCT01590680
Title: An Open Label, Expanded Access Protocol Using 131I-metaiodobenzylguanidine (131I-MIBG) Therapy in Patients With Refractory Neuroblastoma, Pheochromocytoma, or Paraganglioma (Not Eligible for Approved Treatment)
Brief Title: Expanded Access Protocol Using 131I-MIBG
Status: Available | Type: Expanded Access
Sponsor: Jubilant DraxImage Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JDI2007-01
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Neuroblastoma; Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma; Paraganglioma | interventions — 3-Iodobenzylguanidine

INTERVENTIONS:
Radiation: I-131 MIBG — The therapeutic dose (5-18 mCi/kg at investigator's discretion; any dose ≥12 mCi/kg requires stored stem cells) will be diluted in normal saline, and will be infused intravenously over 90-120 minutes.
  Other Names: I-131 Iobenguane; I-131 meta-iodobenzylguanidine

SUMMARY:
Protocol JDI2007-01 is an Expanded Access Protocol with therapeutic 131I-MIBG for patients with neuroblastoma or pheochromocytoma / paraganglioma, who otherwise do not qualify for available treatments, or where approved treatment is not commercially available.

DETAILED DESCRIPTION:
Primary Objectives:

* To provide 131I-MIBG for compassionate use in patients with neuroblastoma, who otherwise do not qualify for inclusion or cannot participate in the sponsor's pivotal Phase II, FDA-approved, clinical trial.
* To provide 131I-MIBG for compassionate use in patients with neuroblastoma in the absence of a commercially available FDA approved product for the indication.
* Provide palliative therapy with 131I-MIBG for patients with advanced neuroblastoma.
* To provide alternative therapeutic 131I-MIBG options for patients with pheochromocytoma / paraganglioma, not qualifying for FDA-approved MIBG treatment.
* To provide alternative therapeutic 131I-MIBG options for patients with pheochromocytoma / paraganglioma, in the absence of a commercially available FDA-approved product for that indication.
* Gain more information about acute and late toxicity of 131I-MIBG therapy for patients with refractory neuroblastoma, pheochromocytoma, or paraganglioma.

Patients will receive a therapeutic dose at the investigator's discretion (5-18 mCi/kg). However, a dose of 12 mCi/kg or higher requires stored stem cells. Patients may be eligible for additional 131I-MIBG treatments (up to a cumulative total of 3 treatments) if they meet certain criteria.

Treatments with 131I-MIBG must be separated by a minimum of six weeks from previous 131I-MIBG therapy. Post-treatment evaluation will be performed 5-9 weeks (35-63 days) post treatment, and patients will be followed every 6 months until 2 years from therapy. All patients will have toxicity monitoring for 2 years following 131I-MIBG therapy, or until going off study.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Diagnosis: Refractory or relapsed neuroblastoma with original diagnosis based on tumor histopathology or elevated urine catecholamines with typical tumor cells in the bone marrow, OR pheochromocytoma or paraganglioma (less than 12 years of age) not amenable to curative surgery.
2. Age ≥12 months and able to cooperate with radiation safety restrictions during therapy period with/without pharmacologic anxiolysis.
3. Disease status: Failure to respond to standard therapy (usually combination chemotherapy with or without radiation and surgery) or development of progressive disease at any time (any new lesion or an increase in size of >25% of a pre-existing lesion). Disease evaluation must be completed within 8 weeks of study entry. If possible, the disease evaluation should take place subsequent to any intervening therapy; if intervening therapy does occur, evaluations should be done as clinically indicated. If patient has received prior treatment with MIBG, they must have a response or stable disease after the most recent MIBG infusion. Patient may have PD after showing an initial response to MIBG therapy (at [or around] the day 35-63 post-MIBG therapy evaluation).
4. Stem cells: Patients must have a hematopoietic stem cell product available for re-infusion after 131I-MIBG treatment at doses of 12 mCi/kg. If no stem cells are available, then the dose of 131I-MIBG should be <12 mCi/kg.
5. Prior Therapy: Patients may enter this study with or without re-induction therapy for recurrent tumor. Patients must have fully recovered from the toxic effects of any prior therapy, meeting the following criteria:

   1. At least 2 weeks should have elapsed since any anti-tumor therapy and the patient must meet certain hematologic criteria.
   2. 3 months should have elapsed in the case of completing external beam radiation for total abdominal, whole lung, total body irradiation (spot irradiation to skull-based metastases is NOT a contraindication). Patients who receive localized emergency radiation to sites of life-threatening or function-threatening disease prior to or immediately after establishment of the definitive diagnosis are not contraindicated for treatment on this protocol.
   3. Cytokine therapy (e.g. G-CSF, GM-CSF, IL-6, erythropoietin) must be discontinued a minimum of 24 hours prior to 131I-MIBG therapy.
   4. Minimum of six weeks from previous 131I-MIBG therapy.
   5. The lifetime cumulative injected activity should be evaluated by the Investigator on a case-by-case basis with special attention to any recovery from past 131I-MIBG dose(s).
   6. For patients who received a stem cell infusion for a previous 131I-MIBG therapy but do NOT have remaining stored stem cells:

   i. If the stem cell reinfusion was protocol driven but not based upon the development of profound cytopenias (e.g. automatic stem cell reinfusion on Day 14), the patient is eligible for retreatment with MIBG at a dose <12 mCi/kg at the investigators discretion; ii. If the stem cell reinfusion was given based upon the development of profound cytopenias, decisions for re-treatment with 131I-MIBG will require a case-by-case evaluation by the Investigator.
6. Organ Function:

   1. Liver function: Bilirubin ≤ 2x upper limit of normal; AST/ALT ≤ 10x upper limit of normal.
   2. Kidney function:

   i. Serum Creatinine ≤ 2x upper limit of normal OR ii. 24-hr creatinine clearance OR GFR ≥ 60 ml/min/1.73m2.

   c. Hematologic Criteria: ANC ≥750/uL; Platelets ≥ 50,000/uL without transfusion if stem cells are not available (ANC ≥ 500 and any platelet count allowed if stem cells available). Patient must be off myeloid growth factors for at least 24 hours. If the patient has received prior treatment with MIBG, they may be thrombocytopenic, but requiring no more than 2 platelet transfusions per week to maintain counts above 20,000/uL. Hemoglobin must be ≥ 10gm/dL (transfusion allowed) regardless of stored stem cell availability.

   d. Normal lung function, as manifested by no dyspnea at rest or exercise intolerance, no oxygen requirement.

   e. No clinically significant cardiac dysfunction.
7. Signed informed consent/assent has been obtained.

EXCLUSION CRITERIA:

1. Patients 12 years and older with iobenguane scan positive, unresectable, locally advanced or metastatic pheochromocytoma or paraganglioma and marketed product is available.
2. Patients eligible for the Phase II (OPTIMUM) trial.
3. Patients with disease of any major organ system that would compromise their ability to withstand therapy. Any significant organ impairment should be discussed with the Principal Investigator prior to patient entry.
4. Because of the teratogenic potential of the study medications, no patients who are pregnant or lactating will be allowed. Patients of childbearing potential, who are sexually active, must practice an effective method of birth control while participating on this study, to avoid possible damage to the fetus . [e.g. intrauterine device, double-barrier method (i.e., diaphragm, or a cervical cap) with intravaginal spermicidal foam, cream or gel], or male partner sterilization throughout the study].
5. Patients who are on hemodialysis
6. Proteinuria, in the absence of urinary infection, within 4 weeks prior to the planned treatment date is a relative contraindication to receiving therapy for patients with pheochromocytoma/paraganglioma. Patients with pheochromocytoma/paraganglioma with any clinically significant proteinuria must have a 24-hr urine protein determination. If proteinuria is confirmed as being above the institutional upper limit of normal, the patient is ineligible for MIBG therapy.
7. Patients with active infections that meet grade 3-4 according to the current version of the NCI CTCAE.
8. Patients with known MIBG-avid parenchymal brain metastases are not eligible. (Patients with leptomeningeal or skull-based metastases are eligible.)

Min Age: 12 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Michigan Medicine, University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - North Carolina Children's Hospital, Chapel Hill, North Carolina
  - Carolinas Medical Center/ Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, American Family Children's Hospital, Madison, Wisconsin